CLINICAL TRIAL: NCT04367155
Title: Efficacy of Tranexamic Acid on Blood Loss During Percutaneous Nephrolithotomy. a Double-blind, Placebo-controlled Randomized Clinical Trial.
Brief Title: Efficacy of Tranexamic Acid on Blood Loss During Percutaneous Nephrolithotomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Diaa Eldin Taha Ramadan Mohamed, Lecturer of urology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS/19.22
Record Dates: First submitted 2020-04-18; First posted 2020-04-29 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Renal Stones; Nephrolithiasis
Keywords: Tranexamic acid; percutanous nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: tranexamic acid during and after percutanous nephrolithotomy procedure
Who Masked: Care Provider, Outcomes Assessor
Masking Description: randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tranexamic acid local (Active Comparator): tranexamic acid inside the irrigation fluid
  Interventions: Drug: Tranexamic acid injection
- tranexamic acid IV (Active Comparator): tranexamic acid injection
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — hemostatics use
  Other Names: tranexamic acid 500 mg

SUMMARY:
Efficacy of tranexamic acid on blood loss during percutaneous nephrolithotomy. a double-blind, placebo-controlled randomized clinical trial.

DETAILED DESCRIPTION:
To evaluate whether intravenous tranexamic acid or tranexamic acid in the irrigation fluid in percutaneous nephrolithotomy (PCNL) in reducing bleeding during and after PCNL.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older
* Stones ≥ 2 cm and/or mild to moderate hydronephrosis.

Exclusion Criteria:

* Age <18 years or Pregnancy
* Bilateral simultaneous PCNL
* Morbid obesity (BMI >40)
* Refuse to complete study requirements
* Untreated UTI
* Atypical bowel interposition by CT
* Tumour in the presumptive access tract area or Potential malignant kidney tumour

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
To assess the value of tranexamic acid | 12 months
  To compare the efficacy and safety of 0.1% IV tranexamic acid versus inside the irrigant fluid tranexamic acid in reducing blood loss during PCNL. Moreover, to assess the adverse events of tranexamic acid.

SECONDARY OUTCOMES:
Hemoglobin drop post PCNL. | 12 months
  Assess fall percentage in hemoglobin drop.
Requirement of blood transfusion post PCNL. | 12 months
  assess the total blood loss and requirement of blood transfusion post PCNL.

CONTACTS AND LOCATIONS:
Overall Officials: Diaa Eldin Taha, MD, Principal Investigator — Lecturer of urology
Locations (1):
- Kafrelsheikh faculty of medicine, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cleveland B, Norling B, Wang H, Gandhi V, Price CL, Borofsky MS, Pais V, Dahm P. Tranexamic acid for percutaneous nephrolithotomy. Cochrane Database Syst Rev. 2023 Oct 26;10(10):CD015122. doi: 10.1002/14651858.CD015122.pub2. PMID 37882229